CLINICAL TRIAL: NCT03841071
Title: Use of the Ostomy Adjustment Scale (OAS) as a Routine Outcome Measure of Adaptation to Life With an Ostomy Along With a Clinical Feedback System in the Follow-up of Ostomy Patients; Does it Promote Adaptation to the Life With an Ostomy?
Brief Title: A Clinical Feedback System in Ostomy Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helse Forde (Other)
Collaborators: Western Norway University of Applied Sciences (Other); Norwegian Nurses Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: 2016255; 2016255 (Other: REC West)
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Ostomy; Quality of Life; Adaptation, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ROM/CFS intervention: The ROM/CFS group (N>100), consists of patients who have undergone urostomy, colostomy, or ileostomy operations, and who are included in the routine follow-up program of the outpatient ostomy clinic at the Department of Surgery, Førde Central Hospital from April 2018 to June 2021.
  Interventions: Other: ROM/CFS intervention

INTERVENTIONS:
Other: ROM/CFS intervention — The intervention (ROM/CFS) includes self-reported measures for adaptation to life with an ostomy and health-related quality of life, as well as patient satisfaction recorded by the clinical feedback system. The measures are electronically assessed before each clinical consultation at 3, 6, and 12 months after surgery, and annually thereafter. The scores are instantly analysed and graphically presented for use during the consultation and the patient and stoma care nurse can discuss the findings.

SUMMARY:
Background: Living with an ostomy can be challenging and adapting to life with an ostomy can be particularly complex, with regard to both the physical and psychosocial aspects. Follow-up with a stoma care nurse is usually performed after surgery to support the adaptation process. In this project, we describe a new model of ostomy care, where a clinical feedback system (CFS) is implemented in order to improve the adaption process of patients with an ostomy. We also present a plan for evaluating patients experience with the CFS and their clinical outcomes.

Methods: We include patients who had recently performed colostomy, ileostomy, or urostomy surgery. The intervention includes self-reported measures for adaptation to life with an ostomy and health-related quality of life (HRQoL), as well as patient experiences and satisfaction recorded by the clinical feedback system. The measures are electronically assessed before each clinical consultation at 3, 6, and 12 months after surgery. The scores are instantly analysed and graphically presented for use during the consultation and the patient and stoma care nurse can discuss the findings. Patient experiences and satisfaction with care will be measured with the Generic Short Patient Experiences Questionnaire. Adaptation to the life with ostomy will be measured with the Ostomy Adjustment Scale, and HRQoL with the Short Form 36.

Discussion: This study presents a novel approach that could lead to improved consultation, more patient involvement, and better adaptation to life with an ostomy.

DETAILED DESCRIPTION:
The study protocol is avaliable on request, and will also be published in a open acsess peer-reviewed journal.

ELIGIBILITY:
Inclusion criteria:

* >18 years of age
* Living with a colostomy, ileostomy, or urostomy for a minimum of 3 months
* Being able to read and write Norwegian

Exclusion criteria:

* < The 3 weeks follow-up after surgery are not included
* Patients who have their ostomy removed <12 months after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone urostomy, colostomy, or ileostomy operations, and who are included in the routine follow-up program at a outpatient ostomy clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
The patient's subjective adaptation to the physical, psychological, and social changes that occur after ostomy surgery | From the 3 months follow-up after surgery to the 12 months follow-up.
  The summary score of the Ostomy Adjustment Scale (lowest possible score is 34 and the highest 204). Higher scores represent better outcomes.

SECONDARY OUTCOMES:
Generic health-related quality of life | From the 3 months follow-up after surgery to the 12 months follow-up.
  The two summary scores of the Short Form-36 (Physical Component Score and Mental Component Score). The lowest possible score is 0 and the highest 100. Higher scores represent better outcomes.

OTHER OUTCOMES:
The patients' satisfaction with the consultation | At the 12 months follow-up after surgery.
  The Session rating scale, using the five item scores seperately (lowest possible score is 0 and the highest 10). Higher scores represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: John R Andersen, PhD, Principal Investigator — Førde Hospital Trust
Locations (1):
- Førde Hospital Trust, Førde, Norway

IPD SHARING:
Plan to Share IPD: Yes
The dataset generated during this study will not be publicly available as the patient consent and approval from the Regional Committee for Medical and Health Research Ethics prevents sharing of individual patient level data in public repositories. However, the data will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from the corresponding author upon reasonable request after publication.
  The study protocol is avaliable on request, and will also be published in a open acsess peer-reviewed journal.
Access Criteria: Supporting information is freely available from The Central Contact Person: Kirsten L Indrebø. Email: kirsten.lerum.indrebo@helse-forde.no.

REFERENCES:
- [Derived] Indrebo KL, Aasprang A, Olsen TE, Andersen JR. Factors associated with leakage in patients with an ostomy: A cross-sectional study. Nurs Open. 2023 Jun;10(6):3635-3645. doi: 10.1002/nop2.1612. Epub 2023 Jan 24. PMID 36691880
- [Derived] Indrebo KL, Aasprang A, Olsen TE, Andersen JR. Psychometric Properties of New Subscales of the Ostomy Adjustment Scale: A Cross-Sectional Study. Patient Relat Outcome Meas. 2021 Mar 15;12:65-75. doi: 10.2147/PROM.S300604. eCollection 2021. PMID 33758568
- [Derived] Indrebo KL, Aasprang A, Olsen TE, Andersen JR. A new model of patient-reported outcome monitoring with a clinical feedback system in ostomy care: rationale, description and evaluation protocol. Health Qual Life Outcomes. 2020 Jan 15;18(1):12. doi: 10.1186/s12955-019-1261-3. PMID 31941516
- See also: Study approval from the Regional Committees for Medical and Health Research Ethics (REC) — https://helseforskning.etikkom.no/prosjekterirek/prosjektregister/prosjekt?_ikbLanguageCode=us